CLINICAL TRIAL: NCT04027530
Title: Phase 4, Randomized, Placebo-controlled, Cross-over Trial to Assess the Effect of 4-week Ertugliflozin (SGLT-2 Inhibitor) Therapy on Renal Oxygenation by BOLD-MRI and Renal Oxygen Consumption by PET Using ¹¹C-acetate in T2DM Without Kidney Disease and Healthy Controls.
Brief Title: Renal Oxygenation, Oxygen Consumption and Hemodynamic Kinetics in Type 2 DIabetes: an Ertugliflozin Study.
Acronym: ROCKIES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, D van Raalte, Dr. D.H. van Raalte, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DC2019 ROCKIES 1
Record Dates: First submitted 2019-07-09; First posted 2019-07-22 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes Mellitus; Diabetic Kidney Disease; Diabetic Nephropathy; Renal Hypoxia; Renoprotection; SGLT2 Inhibitor; Ertugliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — ertugliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ertugliflozin 15mg once daily (Experimental): Once daily treatment with oral ertugliflozin (steglatro) 15mg for 4 consecutive weeks.
  Interventions: Drug: Ertugliflozin 15 mg
- Placebo (Placebo Comparator): Once daily treatment with a placebo pill for 4 consecutive weeks.
  Interventions: Drug: Ertugliflozin 15 mg

INTERVENTIONS:
Drug: Ertugliflozin 15 mg — Once daily treatment with oral ertugliflozin 15mg for 4 consecutive weeks
  Other Names: Steglatro

SUMMARY:
Current study will render insight in to the role of renal hypoxia in the diabetic kidney and is able to associate its finding with measurements of renal perfusion and glomerular filtration rate. Moreover, this research will focus on the effects of sodium-glucose cotransporter 2 inhibition on renal tissue oxygenation and oxygen consumption as well as a change in intrarenal hemodynamics and perfusion, and a shift of fuel metabolites. Elucidation the mechanisms underlying the effects of SGLT2 inhibition will advance our knowledge and contribute to their optimal clinical utilization in the treatment of chronic kidney disease in diabetes and possibly beyond.

DETAILED DESCRIPTION:
Sodium-glucose cotransporter-2 inhibitors (SGLT2-i) are a relatively new class of drugs in the treatment of diabetes and improve glycemic control by blocking SGLT-2 in the proximal tubule, the main transporter of coupled sodium-glucose reabsorption Three large cardiovascular outcome trials (EMPA-REG, CANVAS, DECLARE- TIMI 58) showed SGLT-2 inhibition to have a renoprotective effect, including on renal outcomes. Moreover, the recently publicized CREDENCE trial concluded early after the planned interim analyses showed a striking renoprotective effect of SGLT-2 inhibition in patients with T2DM and CKD. The mechanisms underlying their beneficial effects remain to be elucidated, as the small SGLT-2 induced reduction in glucose level (0.5% HbA1c), bodyweight (about 3%), systolic blood pressure (about 4 mmHg), or uric acid (about 6%) are insufficient to fully account for the effect.

The pathological mechanisms underlying DKD involve complex interactions between metabolic and haemodynamic factors which are not fully understood. However, accumulating evidence of foremost animal studies indicates that a chronic state of renal tissue hypoxia is the final common pathway in the development and progression of diabetic kidney disease. Therefore several hypothesis have been proposed on the alleviation of chronic tissue hypoxia following SGLT-2 inhibition: (1) A decrease in workload by a decrease in GFR. (2) A shift in renal fuel energetics by increasing ketone body oxidation, which renders high ATP/oxygen consumption ratio's compared to glucose or free fatty acids. (3) An improvement of cardiac function and systemic hemodynamics to lead to an increase in renal perfusion, and (4) an increase in erythropoietin (EPO) levels to stimulate oxygen delivery.

Current study will examine the above hypothesis by researching renal oxygenation by BOLD-MRI, oxygen consumption by PET-CT, and hemodynamic kinetics by the Iohexol clearance method/contrast-enhance ultrasound/arterial spin labeling. Blood sampling will allow for the measurement of EPO and ketone bodies, as well as a resting energy expenditure will elucidate a shift in use of energy substrate metabolism. The research will be performed in T2DM without overt kidney disease (n=20) before and after a 4 week treatment with SGLT-2 inhibition (ertugliflozin), and will be compared the obtained results from healthy controls (n=20).

ELIGIBILITY:
Group 1: T2DM patients

Inclusion criteria

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Caucasian*; female or male aged ≥18 years and <80 years. Females must be post-menopausal (defined as no menses >1 year and follicle stimulating hormone (FSH) >31 U/L)*.
* Type 2 diabetes mellitus since at least 3 years with HbA1c ≥ 6.5% (≥57mmol/mol) and <10% (<94mmol/mol)
* An appropriate stable dose of metformin and/or sulfonylurea as glucose-lowering therapy for the last 12 weeks
* Maximum tolerated antihypertensive dose of an ARB for at least 6 weeks prior to randomization.
* eGFR 60-90 ml/min/1.73m²
* BMI 25-35 kg/m² * In order to increase homogeneity

Exclusion criteria

* Involvement in the planning and/or conduction of another study
* Participation in another clinical study with an investigational product during the last 3 months
* Diagnosis of type 1 diabetes mellitus
* CKD defined as eGFR<60 ml/min/1.73m² or albuminuria (defined as an UACR > 2.5 mg/mol).
* Cardiovascular disease event in the last 6 months prior to enrollment as assessed by the investigator, including: myocardial infarction, cardiac surgery or revascularization (CABG/PTCA), unstable angina, heart failure, transient ischemic attack (TIA) or significant cerebrovascular disease, unstable or previously undiagnosed arrhythmia.
* Current/chronic use of the following medication: insulin, thiazolidinediones, GLP-1 receptor agonists, DPP-4 inhibitors, SGLT-2 inhibitors, oral glucocorticoids, non-steroidal anti-inflammatory drugs (NSAIDs), immune suppressants, chemotherapeutics, antipsychotics, tricyclic antidepressants (TCAs), diuretics, and monoamine oxidase inhibitors.
* Current urinary tract infection or active nephritis
* History of ketoacidosis
* History of allergy/hypersensitivity to any of the test agents.

Group 2: Age-matched and eGFR-matched non-diabetic controls Inclusion criteria

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Caucasian*; female or male aged ≥18 years and <80 years. Females must be post-menopausal (defined as no menses >1 year and follicle stimulating hormone (FSH) >31 U/L)*.
* Normal glucose tolerance at screening as confirmed by OGTT
* Maximum tolerated antihypertensive dose of an ARB for at least 6 weeks prior to randomization in case of hypertension.
* BMI 25-35 kg/m2
* eGFR 60-90ml/min * In order to increase homogeneity

Exclusion criteria

* Involvement in the planning and/or conduction of another study
* Participation in another clinical study with an investigational product during the last 3 months
* CKD defined as eGFR<60ml/min or macro-albuminuria or proteinuria
* Cardiovascular disease event in the last 6 months prior to enrollment, as assessed by the investigator, including: myocardial infarction, cardiac surgery or revascularization (CABG/PTCA), unstable angina, heart failure, transient ischemic attack (TIA) or significant cerebrovascular disease, unstable or previously undiagnosed arrhythmia.
* Use of medication that may interfere with study endpoints non-steroidal anti-inflammatory drugs (NSAIDs), immune suppressants, chemotherapeutics, antipsychotics, tricyclic antidepressants (TCAs), diuretics, and monoamine oxidase inhibitors.
* Current urinary tract infection and active nephritis
* Any other condition that prevents participation as judged by investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Renal oxygenation measured by BOLD-MRI (R2*) | After 4 week treatment with ertugliflozin 15mg QD versus placebo
  Renal (separated as cortical and medullar) oxygenation measured by BOLD-MRI (R2*)

SECONDARY OUTCOMES:
Renal oxygen consumption by PET/CT-scan using 11C-Acetate | After 4 week treatment with active drug intervention versus placebo
  Renal oxygen consumption will be measured by PET/CT-scan using 11C-Acetate and compartment model parameter k2
Renal hemodynamics | After 4 week treatment with active drug intervention versus placebo
  GFR and ERPF
Renal efficiency | After 4 week treatment with active drug intervention versus placebo
  Measured as sodium reabsorption divided by oxygen consumption
Cortical blood flow | After 4 week treatment with active drug intervention versus placebo
  measured by contrast-enhanced ultrasound
Renal arterial blood flow | After 4 week treatment with active drug intervention versus placebo
  measured by arterial spin labelling
Acute 24-hour sodium and glucose excretion | After 2 days of treatment with active drug intervention versus placebo
  24-hour sodium and glucose excretion after 2 days
  * Urine osmolality
  * Urinary pH
Chronic 24-hour sodium and glucose excretion | After 4 week treatment with active drug intervention versus placebo
  24-hour sodium and glucose excretion after 4 weeks
Renal tubular function: Urinary pH | After 4 week treatment with active drug intervention versus placebo
  Urinary pH
Renal tubular function: Urine Osmolality | After 4 week treatment with active drug intervention versus placebo
  Urine osmolality
Renal tubular function: sodium transport | After 4 week treatment with active drug intervention versus placebo
  Iohexol corrected sodium excretion
Renal damage markers | After 4 week treatment with active drug intervention versus placebo
  Renal damage markers will include: urinary albumin excretion in 24-hour urine samples and other markers depending on relevant (emerging) metabolic and humoral biomarkers of renal damage, conditional to available budget.
Changes in plasma energy substrate: glucose | After 4 week treatment with active drug intervention versus placebo
  Changes in plasma energy substrate: glucose
Changes in plasma energy substrate: free fatty acids | After 4 week treatment with active drug intervention versus placebo
  Changes in plasma energy substrate: free fatty acids
Changes in plasma energy substrate: ketone bodies | After 4 week treatment with active drug intervention versus placebo
  Changes in plasma energy substrate: ketone bodies
Changes in plasma energy substrate:triglycerides | After 4 week treatment with active drug intervention versus placebo
  Changes in plasma energy substrate:triglycerides
Energy expenditure | After 4 week treatment with active drug intervention versus placebo
  By resting energy expenditure
Changes in erythropoietin (EPO) levels | After 4 week treatment with active drug intervention versus placebo
  Changes in erythropoietin (EPO) levels
Insulin sensitivity | After 4 week treatment with active drug intervention versus placebo
  OGIS and Matsuda Index during an oral glucose tolerance test (OGTT)
Beta-cell function | After 4 week treatment with active drug intervention versus placebo
  Beta-cell function will be derived from HOMA-B modelling during an oral glucose tolerance test (OGTT).
Peripheral insulin extraction | After 4 week treatment with active drug intervention versus placebo
  Arterial-venous difference before and following an OGTT
Total insulin extraction | After 4 week treatment with active drug intervention versus placebo
  Arterial-venous difference before and following an OGTT

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands